CLINICAL TRIAL: NCT00266435
Title: The Usefulness of the HyperQ Stress System in Routine Annual Screening Testing
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-05-3693-ES-CTIL
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Cardiovascular Diseases
Keywords: Asymptomatic subjects; Moderate to high risk for cardiovascular event
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The main objective of this study is to compare the sensitivity and specificity of a new system for analyzing the electrocardiogram (ECG) to the sensitivity and specificity of a conservative treadmill test in asymptomatic subjects, classified by Framingham score as moderate to high risk. Subjects will perform a routine exercise test with the addition of another set of electrodes to record high resolution ECG. All subjects will perform a stress echocardiography. The result of the routine ECG analysis will be compared to the new system and to the echocardiography results.

ELIGIBILITY:
Inclusion Criteria:

* A patient referred to annual screening check
* Classified as being at intermediate or high risk for the development of cardiovascular disease by the Framingham score.
* Signed an Informed Consent Form

Exclusion Criteria:

* A subject who cannot or should not perform an exercise test.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary prevention program
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2005-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Schwammenthal, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel